CLINICAL TRIAL: NCT02185976
Title: Preoperative Anxiety in Paediatric Patients; do Cartoons Help?
Brief Title: Effect of Cartoons on Preoperative Anxiety in Paediatric Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, hafize fisun demir, Assistant Professor, Balikesir University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 2013/051
Record Dates: First submitted 2014-07-04; First posted 2014-07-10 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Anxiety
Keywords: preoperative anxiety; paediatric patients; Cartoon
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cartoon (Active Comparator): paediatric patients undergoing general anesthesia. This group will choose a cartoon movie to watch throughout the preparation until the induction of anesthesia
  Interventions: Other: cartoon
- routine (No Intervention): paediatric patients undergoing general anesthesia

INTERVENTIONS:
Other: cartoon — 5 different cartoons which will be recorded on a tablet PC.
  Arms: cartoon

SUMMARY:
Preoperative Anxiety is a major problem in anesthesia management. Paediatric patients are a special group who need special attention. Some studies have shown that cartoons are a very good tool for distraction in the preoperative period for children.

Our hypothesis is that children watching Cartoons in the preoperative period will have less anxiety and will be fit with preparation.

DETAILED DESCRIPTION:
After local ethics committee approval 60 patients scheduled for various types of surgery will be included.

On the operation day patients are going to be evaluated in the preoperative preparation room. For anxiety evaluation the modified yale preoperative anxiety scale will be used. After this first evaluation patients are going to be separated randomly into two groups; group R (routine) and group C (cartoon). All patients are going to be premedicated with midazolam. The first group will receive their premedication straight after the first evaluation and their response will be recorded as easy, moderate, difficult, does not accept. Group C will choose a cartoon movie (5 different movies are recorded and will be shown through a tablet PC)) and will begin to watch it. After 5 minutes they will receive their premedication and their response will also be recorded. After 30 minutes a physician will try to insert an IV line and the response of the child will also be evaluated and recorded as easy, moderate, difficult and does not allow. Afterwards the patient will be transported into the operation room. In the operation room anesthesia will be induced via Sevoflurane and the response to mask anesthesia will be evaluated with the mask score as it is described before in previous studies. Patients in Group C will continue to watch the cartoon movie until the induction of anesthesia. And the modified yale score will also be reevaluated and recorded.

The family anxiety will be evaluated with the State Trait Anxiety Inventory Scale.

The family and the child will also be interviewed separately, 4 prepared standard questions will be asked in order to understand how the family described the operation.

ELIGIBILITY:
Inclusion Criteria:

* family approval
* age between 3-9
* scheduled for surgery under general anesthesia

Exclusion Criteria:

* history of physiatric disease
* regular medication
* previous history of anesthesia/sedation

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
anxiety score | at the beginning and before induction of anesthesia
  the anxiety score of included patients is going to be evaluated at the beginning in the preparation room and once again in the operation room before induction.

SECONDARY OUTCOMES:
family anxiety scores | Before operation during the first examination
  the anxiety score of the parents is going to be evaluated before the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Hafize Fi Demir, Assist. Prof, Principal Investigator — Balikesir University School of Medicine Department of Anesthesia and Reanimation
Locations (1):
- Balikesir University Faculty of Medicine, Balıkesir, Turkey (Türkiye)